CLINICAL TRIAL: NCT06462092
Title: A Phase I/II Clinical Study of Sacituzumab Govitecan Combined With Intrathecal Chemotherapy for the Treatment of Leptomeningeal Metastases From Her2-negative Breast Cancer
Brief Title: Sacituzumab Govitecan and Intrathecal Chemotherapy for Treating Leptomeningeal Metastases From Her2-negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-027-01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Leptomeningeal Metastases
Keywords: Breast cancer; Her2- (Human Epidermal Growth Factor Receptor 2 Negative); Leptomeningeal Metastases; Sacituzumab Govitecan; Pemetrexed; Intrathecal chemotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis; Breast Neoplasms | interventions — sacituzumab govitecan; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group (Experimental): In the Phase I cohort, a minimum of 3 patients and a maximum of 6 patients were enrolled. If DLT occurred in ≥2 patients, the dose of intrathecal pemetrexed was reduced to 10 mg, and enrollment continued with 6 consecutive patients. If DLT recurred in ≥2 patients, the trial was terminated. if DLT occurred in ≤1 patient, the study advanced to Phase II.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Pemetrexed

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Patients receive Sacituzumab Govitecan 10mg/kg by intravenous infusion on days 1 and 8. Treatment cycles are every 21 days.
  Other Names: Trodelvy
Drug: Pemetrexed — Intrathecal pemetrexed chemotherapy, administered via intracerebroventricular or lumbar puncture, consists of three phases: induction therapy (15 mg twice weekly for 2 weeks), consolidation therapy (once weekly for 4 consecutive weeks), and maintenance therapy (once monthly).
  Other Names: ALIMTA

SUMMARY:
Leptomeningeal metastases (LM) is a lethal complication of malignant tumors, characterized by tumor cell invasion and proliferation within the subarachnoid space. LM from HER2-negative breast cancer remains challenging to treat, with a median overall survival of only 3-6 months despite aggressive therapy. This open-label, uncontrolled Phase I/II clinical study aims to evaluate the safety, feasibility, and potential efficacy of Sacituzumab Govitecan in combination with intrathecal pemetrexed chemotherapy for LM from HER2-negative breast cancer, with the objective of identifying a more effective treatment strategy.

DETAILED DESCRIPTION:
This study is a single-arm, prospective Phase I/II clinical trial, evaluating the safety, feasibility, and potential efficacy of combining Sacituzumab Govitecan with intrathecal pemetrexed chemotherapy for leptomeningeal metastases from HER2-negative breast cancer. The treatment regimen includes intravenous administration of Sacituzumab Govitecan (10 mg/kg) on Days 1 and 8 of each 21-day cycle, continuing until disease progression or unacceptable toxicity. Intrathecal pemetrexed chemotherapy is initiated on Day 2 via intracerebroventricular or lumbar puncture. The treatment is divided into three phases: induction therapy, 15 mg twice weekly for 2 weeks; consolidation therapy, once weekly for 4 weeks; maintenance therapy, once monthly for patients with an effective response until relapse or death. In the Phase I cohort, 3-6 patients were enrolled. If dose-limiting toxicity (DLT) occurred in ≥2 patients, the intrathecal dose of pemetrexed was reduced to 10 mg, and enrollment continued to ensure a total of 6 evaluable patients. If DLT recurred in ≥2 patients among the subsequently enrolled patients, the trial would be terminated. If DLT occurred in ≤1 patient, the trial would proceed to Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. A clear histopathologic diagnosis of breast cancer with HER2-negative subtype (including IHC 0, IHC 1+ or IHC 2+ and ISH negative);
2. Cerebrospinal fluid cytology confirms the presence of leptomeningeal metastases; or imaging findings combined with clinical symptoms and signs are consistent with the diagnosis of leptomeningeal metastases;
3. Age ≥ 18 years old.

Exclusion Criteria:

1. Inadequate organ function: 1) Blood tests: ANC ≤ 1.5 x 10^9/L, PLT ≤ 90 x 10^9/L, Hb ≤ 90 g/L; 2) Blood biochemistry tests: TBIL ≥ 1.5 times the upper limit of normal; 3) ALT and AST ≥ 2.5 times the upper limit of normal;
2. Presence of serious and/or uncontrolled comorbidities that may affect participation: 1) Allergy to study drugs or adjuvant materials; 2) History of immunodeficiency (e.g., HIV-positive or other acquired or congenital immunodeficiency disease); 3) Severe concomitant diseases;
3. Pregnant and breastfeeding female patients; women of childbearing age who are unwilling or unable to use effective contraception;
4. Any other condition that, in the opinion of the investigator, makes the patient ineligible for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose | From the beginning of the treatment until two months after the treatment.
  DLT was defined as Grade 3 neurological toxicities (e.g., chemical meningitis) or any Grade 4 toxicity. If DLT occurred in more than two patients at a given dose level, that dose level was deemed intolerable, and the maximal tolerated dose (MTD) was exceeded. In such cases, an additional three patients were treated at the next lower dose level. The MTD was defined as the dose level at which 0/3 or 1/6 patients experienced DLT, given that at least two patients experiencing DLT at the higher dose.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | From the beginning of the treatment until two months after the treatment.
  The incidence of treatment-related adverse events (AEs) was assessed to determine tolerability and safety. AEs were graded according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03), with Grades 3-5 defined as moderate to severe events.
Clinical response rate | From the beginning of the treatment until two months after the treatment or patient death.
  The Response Assessment in Neuro-Oncology (RANO) criteria for leptomeningeal metastases were used to assess clinical response in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Principal Investigator — Huizhou Hospital of Guangzhou Medical University
Locations (1):
- The Affiliated Huizhou Hospital, Guangzhou Medical University, Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: SAP
Time Frame: Starting 6 months after publication.
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete.

REFERENCES:
- [Background] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065
- [Background] Pan Z, Yang G, He H, Cui J, Li W, Yuan T, Chen K, Jiang T, Gao P, Sun Y, Cong X, Li Z, Wang Y, Pang X, Song Y, Zhao G. Intrathecal pemetrexed combined with involved-field radiotherapy as a first-line intra-CSF therapy for leptomeningeal metastases from solid tumors: a phase I/II study. Ther Adv Med Oncol. 2020 Jul 17;12:1758835920937953. doi: 10.1177/1758835920937953. eCollection 2020. PMID 32733606
- [Background] Rugo HS, Bardia A, Marme F, Cortes J, Schmid P, Loirat D, Tredan O, Ciruelos E, Dalenc F, Gomez Pardo P, Jhaveri KL, Delaney R, Valdez T, Wang H, Motwani M, Yoon OK, Verret W, Tolaney SM. Overall survival with sacituzumab govitecan in hormone receptor-positive and human epidermal growth factor receptor 2-negative metastatic breast cancer (TROPiCS-02): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Oct 21;402(10411):1423-1433. doi: 10.1016/S0140-6736(23)01245-X. Epub 2023 Aug 23. PMID 37633306
- [Background] Bardia A, Hurvitz SA, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Sardesai SD, Kalinsky K, Zelnak AB, Weaver R, Traina T, Dalenc F, Aftimos P, Lynce F, Diab S, Cortes J, O'Shaughnessy J, Dieras V, Ferrario C, Schmid P, Carey LA, Gianni L, Piccart MJ, Loibl S, Goldenberg DM, Hong Q, Olivo MS, Itri LM, Rugo HS; ASCENT Clinical Trial Investigators. Sacituzumab Govitecan in Metastatic Triple-Negative Breast Cancer. N Engl J Med. 2021 Apr 22;384(16):1529-1541. doi: 10.1056/NEJMoa2028485. PMID 33882206